CLINICAL TRIAL: NCT01806896
Title: A Phase 2, Double-blind Randomized, Sequential Treatment Group, Placebo-controlled Study To Evaluate The Safety, Tolerability And Brain Cortico-striatal Function Of 2 Doses Of Pf-02545920 In Subjects With Early Huntington's Disease
Brief Title: Study Evaluating The Safety, Tolerability And Brain Function Of 2 Doses Of PF-0254920 In Subjects With Early Huntington's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A8241016; 2012-004432-31 (EudraCT Number)
Record Dates: First submitted 2013-03-06; First posted 2013-03-07 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2017-12-14 (Actual); Status verified 2017-05

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease | interventions — 2-((4-(1-methyl-4-pyridin-4-yl-1H-pyrazol-3-yl)phenoxy)methyl)quinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 20 mg Arm Cohort A (Experimental)
  Interventions: Drug: PF-02545920
- Placebo Arm Cohort A (Placebo Comparator)
  Interventions: Drug: Placebo
- 5 mg Arm Cohort B (Experimental)
  Interventions: Drug: PF-02545920
- Placebo Arm Cohort B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-02545920 — * Dose will be titrated up every 2 days by 5mg increments: 5mg Days 1-2, 10mg days 3-4, 15mg days 5-6, and reach 20 mg from Days 7 to Day28.
  * Orally, approx. Q12H (range 10-14 hours), administered at least one hour prior to, or two hours after meals.
  * Treatment for 28 days.
  Arms: 20 mg Arm Cohort A
Drug: Placebo — - Orally, approx. Q12H (range 10-14 hours), administered at least one hour prior to, or two hours after meals.
  Dosing for 28 days.
  Arms: Placebo Arm Cohort A
Drug: PF-02545920 — * 5mg dose
  * Orally, approx. Q12H (range 10-14 hours), administered at least one hour prior to, or two hours after meals.
  * Dosing for 28 days.
  Arms: 5 mg Arm Cohort B
Drug: Placebo — * Orally, approx. Q12H (range 10-14 hours), administered at least one hour prior to, or two hours after meals.
  * Dosing for 28 days.
  Arms: Placebo Arm Cohort B

SUMMARY:
This study will evaluate the Safety, Tolerability and Brain Function of 2 doses of PF-0254920 in Subjects with Early Huntington's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of Huntington's Disease
* a CAG repeat expansion equal or great than 39
* a Unified Huntington Disease Rating Scale (UHDRS) Total Motor Score equal or greater than 5 and less than 60
* a UHDRS Total Functional Capacity equal or greater than 9

Exclusion Criteria:

* Subjects with evidence or history of severe acute or chronic medical condition or laboratory abnormality, or significant neurological disorder other than HD.
* Treatment with any antipsychotic medication within 5 weeks of enrollment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Centre d'Investigation Clinique (CIC)/ Institut du Cerveau et de la Möelle Epinière (ICM), Paris, France

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-02545920 20 mg Twice a Day: Participants received PF-02545920 orally every 12 hours according to a titration dosing scheme: 5 mg twice daily (BID) on Days 1-2, 10 mg BID on Days 3-4, 15 mg BID on Days 5-6, and 20 mg BID on Days 7-28; followed by a 7 to 10 day safety evaluation period.
- Placebo Twice a Day: Participants received placebo matched to PF-02545920 orally every 12 hours for 28 days, followed by a 7 to 10 day safety evaluation period.
Period: Overall Study
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Started | 20 | 17
Received Treatment | 19 | 17
Completed | 17 | 17
Not Completed | 3 | 0
Not completed — Adverse Event | 2 | 0
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population included all participants who were randomized and received at least 1 dose of PF-02545920 or placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (12.1) | 43.1 (11.8) | 45.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence without regard to causality in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of treatment and up to the follow-up period that were absent before treatment or that worsened relative to pretreatment state. AEs included both SAEs and non-serious AEs.
Time Frame: Baseline up to Day 38
Population: The safety analysis population included all participants who received at least 1 dose of PF-02545920 or placebo.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  AEs | 18 | 14
  SAEs | 1 | 1

2. Primary Outcome: Number of Participants With Laboratory Abnormalities Meeting the Criteria for Potential Clinical Concern (Without Regard to Baseline Abnormality)
Description: The following laboratory parameters were analyzed: hematology (hemoglobin, hematocrit, red blood cell [RBC] count, platelet count, white blood cell [WBC] count, total neutrophils, eosinophils, monocytes, basophils, lymphocytes); blood chemistry (blood urea nitrogen [BUN], creatinine, glucose, calcium, sodium, potassium, chloride, total bicarbonate, aspartate aminotransferase [AST], alanine aminotransferase [ALT], total and direct bilirubin, alkaline phosphatase, uric acid, albumin, and total protein; urinalysis (pH, glucose, protein/albumin, hemoglobin/blood, ketones/acetone, nitrites, leukocyte esterase, microscopy [if urine dipstick was positive for blood, protein, nitrites or leukocyte esterase]); others (urine/serum pregnancy test, glycosylated hemoglobin [HbA1c, if diabetic]).
Time Frame: Baseline up to Day 38
Population: The safety analysis population included all participants who received at least 1 dose of PF-02545920 or placebo.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants | 8 | 8

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs assessment included pulse rate and blood pressure. Criteria for vital sign values meeting potential clinical concern included: supine/sitting pulse rate less than (<)40 or greater than (>)120 beats per minute (bpm), standing pulse rate <40 or >140 bpm; systolic blood pressure (SBP) of greater than or equal to (>=)30 millimeters of mercury (mmHg) change from baseline or SBP <90 mmHg, diastolic blood pressure (DBP) >=20 mmHg change from baseline or DBP <50 mmHg.
Time Frame: Baseline up to Day 38
Population: The safety analysis population included all participants who received at least 1 dose of PF-02545920 or placebo.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  Supine SBP <90 mmHg | 0 | 0
  Standing SBP <90 mmHg | 1 | 0
  Supine DBP <50 mmHg | 2 | 1
  Standing DBP <50 mmHg | 1 | 0
  Supine Pulse Rate <40 or >120 bpm | 0 | 0
  Standing Pulse Rate <40 or >140 bpm | 1 | 0
  Increase From Baseline in Supine SBP >=30 mmHg | 1 | 0
  Increase From Baseline in Standing SBP >=30 mmHg | 2 | 2
  Increase From Baseline in Supine DBP >=20 mmHg | 1 | 0
  Increase From Baseline in Standing DBP >=20 mmHg | 1 | 0
  Decrease From Baseline in Supine SBP >=30 mmHg | 1 | 0
  Decrease From Baseline in Standing SBP >=30 mmHg | 1 | 0
  Decrease From Baseline in Supine DBP >=20 mmHg | 2 | 1
  Decrease From Baseline in Standing DBP >=20 mmHg | 3 | 0

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG parameters included PR interval, QRS complex, and corrected QT interval using Fridericia's formula (QTcF). Criteria for ECG changes meeting potential clinical concern included: PR interval ≥200 milliseconds (msec) or ≥25% increase when baseline is >100 msec; QRS interval ≥50% increase from baseline when baseline is less than or equal to (<=)200 msec; and QTcF ≥450 msec or ≥30 msec increase from baseline.
Time Frame: Baseline up to Day 38
Population: The safety analysis population included all participants who received at least 1 dose of PF-02545920 or placebo.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  PR Interval >=200 msec | 1 | 1
  PR Interval >=300 msec | 0 | 0
  QTcF Interval 450-<480 msec | 2 | 0
  QTcF Interval 480-<500 msec | 0 | 0
  QTcF Interval >=500 msec | 0 | 0
  PR Interval >=25% increase when baseline >100 msec | 0 | 0
  PR Interval >=25% increase when baseline >200 msec | 0 | 0
  QRS >=50% increase when baseline <=100 msec | 0 | 0
  QRS >=50% increase when baseline <=200 msec | 0 | 0
  QTcF Interval Increase 30-<60 msec | 1 | 0
  QTcF Interval Increase >=60 msec | 0 | 0

5. Primary Outcome: Number of Participants With Change From Baseline in Body Weight of >=7%
Description: Weight assessment was performed by a study physician or a trained study nurse and was included in the physical examination.
Time Frame: Baseline up to Day 38
Population: The safety analysis population included all participants who received at least 1 dose of PF-02545920 or placebo.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants | 0 | 0

6. Primary Outcome: Categorical Summary of Participants Meeting Stopping Criteria
Description: Absolute neutrophil count (ANC) and WBC were monitored for safety. Participants with WBC <3000 but >=2000 cells/mm^3 or ANC <1500 but >=1000 cells/mm^3 were to have study treatment suspended. Participants with WBC <2000 or ANC <1000 cells/mm^3 were to be discontinued from study participation.
Time Frame: Baseline up to Day 38
Population: The safety analysis population included all participants who received at least 1 dose of PF-02545920 or placebo.
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  WBC 2000-3000 or ANC 1000-1500 cells/mm^3 | 0 | 1
  WBC <2000 or ANC <1000 cells/mm^3 | 0 | 0
  Discontinued/Suspended Due to WBC or ANC Findings | 0 | 0
  ANC<500 cells/mm^3 | 0 | 0

7. Primary Outcome: Change From Baseline in Unified Huntington Disease Rating Scale (UHDRS) Total Motor Score at Day 28
Description: The UHDRS is a clinical rating scale to provide a uniform assessment of the clinical features and course of Huntington Disease. The Total Motor Score (TMS) is 1 of the 6 components of UHDRS, includes 31 items, and ranges from a scale of 0 to 124 (higher scores indicate more severe disease).
Time Frame: Baseline, Day 28
Population: The full analysis population included all participants randomized and had taken at least 1 dose of PF-02545920 or placebo.
Measure: Least Squares Mean (90% Confidence Interval); unit: units on a scale
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
units on a scale | 0.19 (6.23) [-1.73 to 2.12] | 0.90 (5.70) [-1.14 to 2.94]
Statistical Analysis 1: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Day 28); Test type: Superiority or Other; p = 0.68, ANCOVA — 2-sided p-value; Treatment differences are based on a mixed effect model including treatment as fixed effects and baseline, age, gender and CAG repeats as covariates; Mean Difference (Final Values) = -0.71, 90% CI 2-sided [-3.56 to 2.15], Standard Error of Mean 1.68

8. Primary Outcome: Number of Participants With Suicidal Tendencies (C-SSRS Mapped to C-CASA) at Baseline
Description: C-SSRS is a participant rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses), and intensity of ideation (rated 1=low severity to 5=high severity). Yes/No responses are mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories: completed suicide, suicide attempt, preparatory acts towards imminent suicidal behavior, suicidal ideation, and self-injurious behavior, or no suicidal intent. A participant could have a yes or no response in more than 1 category.
Time Frame: Baseline (Day 1)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  Completed Suicide | 0 | 0
  Suicide Attempt | 0 | 0
  Acts Towards Imminent Suicidal Behavior | 0 | 0
  Suicidal Ideation | 1 | 0
  Self-Injurious Behavior, No Suicidal Intent | 0 | 0

9. Secondary Outcome: Change From Baseline in Functional Magnetic Resonance Imaging (fMRI) in Monetary Incentive Delay (MID) Task at Day 28
Description: The monetary incentive delay (MID) task is established as a reliable method to elicit ventral striatal (VS) activity in relation to reward/punishment anticipation and tracked with dysfunctionalities across a range of conditions in which incentive motivation is thought to be abnormal (schizophrenia, depression, substance abuse, and pathological gambling). Pharmacological intervention has demonstrated reversal of observed deficit. The beta contrast value of 'REW' is for analysis of reward-related activity in VS within the task-related 'reward network' during the gain condition (relative to neutral) of the MID task. The changes in beta contrasts (fMRI) provided are changes in parameter estimates and do not have a unit of measure.
Time Frame: Baseline (Day 1), Day 28
Population: The analysis population included all participants randomized, who had taken at least 1 dose of PF-02545920 or placebo and who had valid data (thresholded by acceptable motion). n=number of participants analyzed in the respective arms. The per-protocol set (PPS) table was used, not the full analysis set (FAS) table.
Measure: Least Squares Mean (90% Confidence Interval); unit: beta contrasts
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 10 | 12
beta contrasts
  Cue Rew>Neut Left VS | 0.01 (1.15) [-0.43 to 0.45] | 0.11 (1.13) [-0.29 to 0.50]
  Cue Rew>Neut Right VS | -0.20 (1.11) [-0.66 to 0.26] | -0.05 (1.32) [-0.47 to 0.37]
  Out_win_Rew>Out_win N Left VS | 0.20 (2.33) [-0.26 to 0.66] | 0.45 (1.13) [0.03 to 0.87]
  Out_win_Rew>Out_win N Right VS | 0.36 (2.00) [-0.04 to 0.77] | 0.89 (1.14) [0.53 to 1.26]
Statistical Analysis 1: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Cue Rew>Neut Left VS); Test type: Superiority or Other; p = 0.79, ANCOVA — 2-sided p-value; Treatment differences are based on a mixed effect model including treatment as fixed effect and baseline, age, gender and CAG repeats as covariates; Least square mean = -0.10, 90% CI 2-sided [-0.72 to 0.52], Standard Error of Mean 0.36
Statistical Analysis 2: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Cue Rew>Neut Right VS); Test type: Superiority or Other; p = 0.70, ANCOVA — 2-sided p-value; [statistical method as in outcome 9, analysis 1]; Least square mean = -0.15, 90% CI 2-sided [-0.80 to 0.51], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Out_win_Rew>Out_win N Left VS); Test type: Superiority or Other; p = 0.51, ANCOVA — 2-sided p-value; [statistical method as in outcome 9, analysis 1]; Least square mean = -0.25, 90% CI 2-sided [-0.89 to 0.40], Standard Error of Mean 0.37
Statistical Analysis 4: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Out_win_Rew>Out_win N Right VS); Test type: Superiority or Other; p = 0.13, ANCOVA — 2-sided p-value; [statistical method as in outcome 9, analysis 1]; Least square mean = -0.53, 90% CI 2-sided [-1.10 to 0.04], Standard Error of Mean 0.33

10. Primary Outcome: Number of Participants With Suicidal Tendencies (C-SSRS Mapped to C-CASA) at Day 7
Description: C-SSRS is a participant rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses), and intensity of ideation (rated 1=low severity to 5=high severity). Yes/No responses are mapped to Columbia Classification Algorithm of Suicide Assessment (C-CASA) categories: completed suicide, suicide attempt, preparatory acts toward imminent suicidal behavior, suicidal ideation, and self-injurious behavior, or no suicidal intent. A participant could have a yes or no response in more than 1 category.
Time Frame: Day 7
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  Completed Suicide | 0 | 0
  Suicide Attempt | 0 | 0
  Acts Towards Imminent Suicidal Behavior | 0 | 0
  Suicidal Ideation | 0 | 0
  Self-Injurious Behavior, No Suicidal Intent | 0 | 0

11. Primary Outcome: Number of Participants With Suicidal Tendencies (C-SSRS Mapped to C-CASA) at Day 28
Description: as for outcome 10
Time Frame: Day 28
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 19 | 17
participants
  Completed Suicide | 0 | 0
  Suicide Attempt | 0 | 0
  Acts Towards Imminent Suicidal Behavior | 0 | 0
  Suicidal Ideation | 2 | 0
  Self-Injurious Behavior, No Suicidal Intent | 0 | 0

12. Secondary Outcome: Change From Baseline in Grip Strength Incentive Motivation Task at Day 28: Percent of Maximum Voluntary Contraction (MVC)
Description: This incentive force task was developed to independently dissociate the degree to which a participant responds to reward motivation versus emotional motivation. The task itself included 12 repetitions of 9 trial types, for a total of 108 trials, grouped in a single session lasting about 20 minutes. The trial types were generated according to a combination of 3 emotional categories (negative, neutral, and positive pictures presented) and to 3 monetary incentives (0.01, 0.1, and 1€). Emotional categories and monetary incentives were randomly distributed over the trials and the sequence was fixed such that all subjects were assessed on the exact same task. For each trial, the subject was first presented with an emotional picture displayed on screen for 3000 milliseconds (ms).
Time Frame: Baseline, Day 28
Population: The analysis population included all participants randomized, who had taken at least 1 dose of PF-02545920 or placebo and who had valid data (acceptable task engagement). n=number of participants analyzed in the respective arms. The PPS table was used, not the FAS table.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage of MVC
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Number analyzed (Participants) | 16 | 17
percentage of MVC
  Neutral Emotional Incentive Day 28 | 0.93 [-3.28 to 5.14] | -6.37 [-10.43 to -2.31]
  Positive Emotional Incentive Day 28 | 1.10 [-3.10 to 5.31] | -6.47 [-10.53 to -2.40]
  Negative Emotional Incentive Day 28 | 0.18 [-4.02 to 4.39] | -7.10 [-11.16 to -3.04]
  0.01 Euro Monetary Incentive Day 28 | -13.47 [-17.79 to -9.14] | -14.45 [-18.59 to -10.31]
  0.1 Euro Monetary Incentive Day 28 | -1.19 [-5.43 to 3.06] | -5.97 [-10.04 to -1.89]
  1 Euro Monetary Incentive Day 28 | 16.85 [12.49 to 21.21] | 0.50 [-3.78 to 4.78]
Statistical Analysis 1: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Emotional Incentive-Neutral) Day 28; Test type: Superiority or Other; p = 0.04, ANCOVA — 2-sided p-value; Mixed effect model including treatment, incentive and treatment*incentive as fixed effects; baseline, age, gender and CAG repeats as covariates; Least square mean = 7.30, 90% CI 2-sided [1.43 to 13.18], Standard Error of Mean 3.57
Statistical Analysis 2: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Emotional Incentive-Positive) Day 28; Test type: Superiority or Other; p = 0.03, ANCOVA — 2-sided p-value; [statistical method as in outcome 12, analysis 1]; Least square mean = 7.57, 90% CI 2-sided [1.69 to 13.45], Standard Error of Mean 3.57
Statistical Analysis 3: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Emotional Incentive-Negative) Day 28; Test type: Superiority or Other; p = 0.04, ANCOVA — 2-sided p-value; [statistical method as in outcome 12, analysis 1]; Least square mean = 7.28, 90% CI 2-sided [1.41 to 13.15], Standard Error of Mean 3.56
Statistical Analysis 4: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Monetary Incentive-0.01 Euro) Day 28; Test type: Superiority or Other; p = 0.78, ANCOVA — 2-sided p-value; [statistical method as in outcome 12, analysis 1]; Least square mean = 0.98, 90% CI 2-sided [-4.91 to 6.87], Standard Error of Mean 3.58
Statistical Analysis 5: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Monetary Incentive-0.1 Euro) Day 28; Test type: Superiority or Other; p = 0.18, ANCOVA — 2-sided p-value; [statistical method as in outcome 12, analysis 1]; Least square mean = 4.78, 90% CI 2-sided [-1.11 to 10.67], Standard Error of Mean 3.58
Statistical Analysis 6: Comparison: PF-02545920 20 mg Twice a Day vs Placebo Twice a Day; PF-02545920 versus Placebo (Monetary Incentive-1 Euro) Day 28; Test type: Superiority or Other; p < 0.01, ANCOVA — 2-sided p-value; [statistical method as in outcome 12, analysis 1]; Least square mean = 16.35, 90% CI 2-sided [10.46 to 22.24], Standard Error of Mean 3.58

ADVERSE EVENTS:
Time Frame: Baseline up to Day 38
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | PF-02545920 20 mg Twice a Day | Placebo Twice a Day
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/17
Other Adverse Events (participants affected / at risk) | 18/19 | 14/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 20 mg Twice a Day (N=19) | Placebo Twice a Day (N=17)
Chorea (Nervous system disorders) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-02545920 20 mg Twice a Day (N=19) | Placebo Twice a Day (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Palpitations (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2
Dry mouth (Gastrointestinal disorders) | 4 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 2 | 1
Fatigue (General disorders) | 8 | 4
Feeling hot (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Thirst (General disorders) | 1 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Electrocardiogram QRS complex prolonged (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Akathisia (Nervous system disorders) | 2 | 0
Chorea (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 6
Migraine (Nervous system disorders) | 1 | 1
Oromandibular dystonia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 3 | 0
Aggression (Psychiatric disorders) | 1 | 0
Bradyphrenia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Irritability (Psychiatric disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Negative thoughts (Psychiatric disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 0
Hot flush (Vascular disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
The study was initially designed to include 20 mg BID and 5 mg BID. Interim analysis of 20 mg BID/placebo supported the development of PF-02545920, and therefore, 5 mg BID was not enrolled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.